CLINICAL TRIAL: NCT02187445
Title: Inhaled Corticosteroid Use to Prevent Acute Chest Syndrome Recurrence in Children Between 1 and 4 With Sickle Cell Disease: a Feasibility Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Emory University (Other); Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Michael DeBaun, Professor of Pediatrics and Medicine, Vice Chair of Clinical Research in Pediatrics, JC Peterson Endowed Chair in Pediatrics, Director, Vanderbilt-Meharry Center of Excellence in Sickle Cell Disease, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DDCF2014086
Record Dates: First submitted 2014-06-27; First posted 2014-07-11 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Sickle Cell Disease; Asthma; Acute Chest Syndrome
Keywords: Sickle Cell Disease; Budesonide inhalation suspension; Acute Chest Syndrome
MeSH Terms: conditions — Anemia, Sickle Cell; Asthma; Acute Chest Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Budesonide inhalation suspension (Experimental): To determine the acceptability of budesonide inhalation suspension (BIS) 0.5 QD for 6 months for children with SCD that develop ACS between 1 and 4 years of age (n=10).
  Interventions: Drug: Budesonide inhalation suspension

INTERVENTIONS:
Drug: Budesonide inhalation suspension — To determine the acceptability of budesonide inhalation suspension (BIS) 0.5 QD for 6 months for children with SCD that develop ACS between 1 and 4 years of age (n=10).
  Other Names: inhaled corticosteroids

SUMMARY:
Acute and chronic pulmonary complications with concomitant inflammatory response are a leading cause of morbidity and mortality in children with sickle cell disease (SCD). Acute chest syndrome (ACS), defined broadly as an increase in respiratory effort, fever and new radiodensity on chest x-ray, is a major cause of death in children and adults with SCD. There is a high rate of ACS in children between 1 and 4 years of age that is associated with an asthma diagnosis, and children with ACS events before 4 years of age have a 50% rate of being hospitalized for either ACS or pain within 1 year of admission. For children with SCD that develop ACS, the investigators propose that the use of budesonide inhalation suspension (BIS) will attenuate pulmonary inflammation after an ACS episode and will decrease future vaso-occlusive pain and ACS episodes. Through a single-arm prospective feasibility trial and in preparation for a limited-institution randomized trial, the investigators plan to test the following primary hypothesis for a phase III definitive trial: In children with SCD admitted to the hospital for an ACS episode between 1 and 4 years of age, low dose BIS for 6 months will result in a 50% reduction in the recurrent incidence rate of ACS or pain requiring hospitalization. Through this trial, the investigators will determine the acceptability of and adherence to BIS in the study population. The investigators will track respiratory symptoms in cases versus controls over 6 months. Finally, the investigators will explore the impact of BIS on biological correlates (sVCAM-1).

ELIGIBILITY:
Inclusion Criteria:

* 1) confirmed diagnosis of sickle cell disease (SCD)
* 2) age between 1 and 4 years (must have reached 1st but not yet 4th birthday)
* 3) a prior diagnosis of ACS, defined as acute respiratory illness with a new radiodensity on CXR, and one of the following: fever (temperature > 38.50C), decrease in oxygen saturation more than 3% from baseline, or increase in respiratory rate above baseline

Exclusion Criteria:

* 1) patients already taking inhaled corticosteroids
* 2) those receiving blood transfusions for elevated TCD or strokes
* 3) presents over 2 weeks after discharge from hospital following initial ACS episode.

Participants may be on hydroxyurea and participate in this trial.

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2017-02-13 (Actual)

PRIMARY OUTCOMES:
The acceptability of budesonide inhalation suspension | 6 Months
  Specific Aim 1: To determine the acceptability of budesonide inhalation suspension (BIS) 0.5 QD for 6 months for children with SCD that develop ACS between 1 and 4 years of age (n=10). We will determine the proportions of eligible families who were willing to participate and families that enrolled and elected to stay throughout the six months of the trial. We will also assess adherence to BIS using the Morisky scale; this will be our primary outcome. If the participation rate for the trial is less than 60%, the dropout rate is greater than 20%, or if our adherence rate is poor as measured by the Morisky scale, then alternative strategies for recruitment, retention and adherence must be considered.

SECONDARY OUTCOMES:
The impact of BIS on biological correlates of inflammation. | 12 weeks (or between 8-16 weeks) and at 24 weeks (or between 20-28 weeks)
  Specific Aim 2: To explore the impact of BIS on biological correlates of inflammation. For this purpose, a blood sample measurement will be taken at baseline, at 12 weeks (between 8-16 weeks) and at 24 weeks (between 20-28 weeks), as per routine clinic visits. The research visit will be coordinated with the standard care visits and phlebotomy. Soluble vascular cell adhesion molecule-1 (sVCAM-1), a marker of chronic vasculopathy, will be the primary measure of vascular injury. Secondary outcome measures will include additional inflammatory markers (sP-selectin, sE-selectin, IL-1B, IL-6, TNFα, IFN-y, leukotrienes).

OTHER OUTCOMES:
Quality of life for guardians of children with sickle cell disease and ACS | 0 weeks, 12 weeks (or between 8-16 weeks) and at 24 weeks (or between 20-28 weeks)
  At each clinic visit, we will also collect patient-centered outcomes, assessing caregiver burden. Data will be collected using the Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ), validated for parents of children with asthma.
Respiratory symptoms | 6 months, monthly
  Using the TRACK survey, validated for guardians of children under the age of 5 years, we will call families monthly to collect data on respiratory symptoms over the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R DeBaun, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States